CLINICAL TRIAL: NCT00267657
Title: Assessment of Interactions Between IV Methamphetamine and Reserpine
Brief Title: A Phase 1 Parallel-Group, Double-Blind, Placebo-Controlled Cardiovascular and Behavioral Study Assessing Interactions Between Single Doses of Oral Reserpine and Intravenous Methamphetamine - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-0006-1
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-12

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Reserpine

INTERVENTIONS:
Drug: Reserpine

SUMMARY:
In this parallel group clinical pharmacology laboratory experiment, we will assess pharmacodynamic interactions (with a focus on cardiovascular effects) of a 15 mg intravenous methamphetamine dose and single oral doses of reserpine (0.5 and 1.0 mg) or placebo.

DETAILED DESCRIPTION:
In this parallel group clinical pharmacology laboratory experiment, we will assess pharmacodynamic interactions (with a focus on cardiovascular effects) of a 15 mg intravenous methamphetamine dose and single oral doses of reserpine (0.5 and 1.0 mg) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Please contact site for more details

Exclusion Criteria:

* Please contact site for more details

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2004-11

PRIMARY OUTCOMES:
Craving
Cardiovascular
Subjective symptoms/Mood Effects
CNS norepinephrine turnover

CONTACTS AND LOCATIONS:
Overall Officials: Reese Jones, M.D., Principal Investigator — Langley Porter Psychiatric Institute
Locations (1):
- U of CA, San Francisco, San Francisco, California, United States